CLINICAL TRIAL: NCT04103567
Title: Determination of Microbiological Factors Associated With Poor Response to Neoadjuvant Therapy in Rectal Cancers: Focus on Cyclomodulin-producing Escherichia Coli
Brief Title: Determination of Microbiological Factors Associated With Poor Response to Neoadjuvant Treatment in Rectal Cancers
Acronym: MICARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2019-14-MIR
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
Keywords: rectal; cancer; cyclomodulin; microbiological factors
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): Fecal samples collected at different times : During inclusion consultation with surgeon, after neoadjuvant treatment and before surgery,
  In parallel to this fecal collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — Fecal samples collected at different times : during inclusion consultation with surgeon, after neoadjuvant treatment and before surgery.

SUMMARY:
The objective of this project is to determine in a non-invasive manner (fecal samples) the predictive value of the intestinal microbiota and the presence of genotoxin-producing bacteria on the response to neoadjuvant treatment in rectal cancer. This could lead to a better understanding and selection of patients for personalized treatment in rectal cancer.

DETAILED DESCRIPTION:
Rectal cancer is the 8th leading cause of cancer in the world with more than 300,000 deaths in 2018. In addition to surgery, neoadjuvant treatment has proven its value in reducing local recurrences. Evaluation of the response to neoadjuvant treatment (essential for the subsequent therapeutic decision but also for the oncological prognosis. It is based on rectal magnetic resonance imaging, completed after surgery by anatomopathology. A personalised treatment with therapeutic de-escalation or intensification for aggressive tumours can be decided depending on the response to Neoadjuvant treatment. Thus, knowledge of the predictive factors of response to neoadjuvant treatment would permit to anticipate and adapt care.

The intestinal microbiota is a true microbial organ, playing a major role in maintaining intestinal homeostasis. Some bacterial species have been identified and suspected of playing a role in colorectal carcinogenesis. Among these species, genotoxin-producing Escherichia coli (CPEC) strains such as colibactin (cyclomodulin encoded by the genomic islet pks) are preferentially detected in patients with colorectal cancer (CRC), especially the most aggressive forms. Recent studies show that the intestinal microbiota is a prognostic factor in the response to certain chemotherapies or immunotherapies, but little work has been done on its potential influence on the effectiveness of radiotherapy. This suggests the possibility of using these biomarkers associated with response to neoadjuvant treatment.

The objective of this project is to determine in a non-invasive manner (fecal samples) the predictive value of the intestinal microbiota and the presence of genotoxin-producing bacteria on the response to neoadjuvant treatment in rectal cancer. This could lead to a better understanding and selection of patients for tailored treatment in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven lower and mid-rectal adenocarcinoma at clinical stage II and III
2. Patient is to receive neoadjuvant treatment (radiochemotherapy or chemotherapy or radiotherapy). Induction chemotherapy such as folfox or folfirinox is allowed
3. Patient who has signed the informed consent of the study
4. Male or female ≥ 18 years old
5. Appropriate contraceptive measures should be used by both men and non-menopausal women before entering the trial until at least 8 weeks after the last course of radiochemotherapy. The investigator should inform the patient about the contraceptive measures to be used.

Exclusion Criteria:

1. Antibiotic treatment at the time or in the month preceding stool sampling
2. Presence of an ostomy
3. Previous treatment for rectal cancer
4. Patient not affiliated to a French social protection system
5. Patient not in favour of good compliance with treatment for psychological, family, social or geographical reasons
6. Legal incapacity (Patient under curatorship or guardianship)
7. Prior radiation therapy or pelvic curia in the year prior to inclusion
8. History of other cancers in the last 5 years (except for in-situ cervical carcinomas and non-melanoma skin carcinomas treated optimally)
9. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
The ratio between the proportions of poor response to neoadjuvant treatment in populations so-called "exposed" (patients colonized by bacteria producing toxins (cyclomodulin) and unexposed (patients not colonized by bacteria producing toxins) | About 1 years

SECONDARY OUTCOMES:
Change of cyclomodulin-Producing Escherichia Coli colonization rate before and after neoadjuvant treatment | About 1 years
Change of cyclomodulin-Producing Escherichia Coli prevalence before and after neoadjuvant treatment | About 1 years
Change of prevalence forming the overall bacterial composition before and after neoadjuvant treatment | About 1 years
Change of colonization rate (in addition to cyclomodulin-Producing Escherichia Coli) forming the overall bacterial composition before and after neoadjuvant treatment | About 1 years
Relative risk of poor response to neoadjuvant treatment in colonized patients with other bacteria ("exposed") compared to non-colonized patients ("unexposed") | About 1 years
Proportion of patients colonized according to the modality of the clinical variable age | About 1 years
Proportion of patients colonized according to the modality of the clinical variable gender | About 1 years
Proportion of patients colonized according to the modality of the clinical variable body mass index | About 1 years
Overall survival in colonized people by the different types of bacteria that form the overall bacterial composition (including cyclomodulin-Producing Escherichia Coli) compared to non-colonized people | About 1 years
Disease-free survival in colonized people by the different types of bacteria that form the overall bacterial composition (including cyclomodulin-Producing Escherichia Coli) compared to non-colonized people | About 1 years
Specific survival in colonized people by the different types of bacteria that form the overall bacterial composition (including cyclomodulin-Producing Escherichia Coli) compared to non-colonized people | About 1 years
Types of other bacteria forming the overall bacterial composition before neoadjuvant treatment | About 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUANET, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (2):
- France (2):
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy De Dôme

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Gerard JP, Andre T, Bibeau F, Conroy T, Legoux JL, Portier G, Bosset JF, Cadiot G, Bouche O, Bedenne L; Societe Francaise de Chirurgie Digestive (SFCD), Societe Francaise d'Endoscopie Digestive (SFED0), Societe Francaise de Radiotherapie Oncologique (SFRO). Rectal cancer: French Intergroup clinical practice guidelines for diagnosis, treatments and follow-up (SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO). Dig Liver Dis. 2017 Apr;49(4):359-367. doi: 10.1016/j.dld.2017.01.152. Epub 2017 Jan 20. PMID 28179091
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Dworak O, Keilholz L, Hoffmann A. Pathological features of rectal cancer after preoperative radiochemotherapy. Int J Colorectal Dis. 1997;12(1):19-23. doi: 10.1007/s003840050072. PMID 9112145
- [Background] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Background] Renehan AG, Malcomson L, Emsley R, Gollins S, Maw A, Myint AS, Rooney PS, Susnerwala S, Blower A, Saunders MP, Wilson MS, Scott N, O'Dwyer ST. Watch-and-wait approach versus surgical resection after chemoradiotherapy for patients with rectal cancer (the OnCoRe project): a propensity-score matched cohort analysis. Lancet Oncol. 2016 Feb;17(2):174-183. doi: 10.1016/S1470-2045(15)00467-2. Epub 2015 Dec 17. PMID 26705854
- [Background] Rullier E, Rouanet P, Tuech JJ, Valverde A, Lelong B, Rivoire M, Faucheron JL, Jafari M, Portier G, Meunier B, Sileznieff I, Prudhomme M, Marchal F, Pocard M, Pezet D, Rullier A, Vendrely V, Denost Q, Asselineau J, Doussau A. Organ preservation for rectal cancer (GRECCAR 2): a prospective, randomised, open-label, multicentre, phase 3 trial. Lancet. 2017 Jul 29;390(10093):469-479. doi: 10.1016/S0140-6736(17)31056-5. Epub 2017 Jun 7. PMID 28601342
- [Background] Rouanet P, Rullier E, Lelong B, Maingon P, Tuech JJ, Pezet D, Castan F, Nougaret S; and the GRECCAR Study Group. Tailored Treatment Strategy for Locally Advanced Rectal Carcinoma Based on the Tumor Response to Induction Chemotherapy: Preliminary Results of the French Phase II Multicenter GRECCAR4 Trial. Dis Colon Rectum. 2017 Jul;60(7):653-663. doi: 10.1097/DCR.0000000000000849. PMID 28594714
- [Background] Savage DC. Microbial ecology of the gastrointestinal tract. Annu Rev Microbiol. 1977;31:107-33. doi: 10.1146/annurev.mi.31.100177.000543. No abstract available. PMID 334036
- [Background] Nougayrede JP, Taieb F, De Rycke J, Oswald E. Cyclomodulins: bacterial effectors that modulate the eukaryotic cell cycle. Trends Microbiol. 2005 Mar;13(3):103-10. doi: 10.1016/j.tim.2005.01.002. PMID 15737728
- [Background] Nougayrede JP, Homburg S, Taieb F, Boury M, Brzuszkiewicz E, Gottschalk G, Buchrieser C, Hacker J, Dobrindt U, Oswald E. Escherichia coli induces DNA double-strand breaks in eukaryotic cells. Science. 2006 Aug 11;313(5788):848-51. doi: 10.1126/science.1127059. PMID 16902142
- [Background] Bonnet M, Buc E, Sauvanet P, Darcha C, Dubois D, Pereira B, Dechelotte P, Bonnet R, Pezet D, Darfeuille-Michaud A. Colonization of the human gut by E. coli and colorectal cancer risk. Clin Cancer Res. 2014 Feb 15;20(4):859-67. doi: 10.1158/1078-0432.CCR-13-1343. Epub 2013 Dec 13. PMID 24334760
- [Background] Buc E, Dubois D, Sauvanet P, Raisch J, Delmas J, Darfeuille-Michaud A, Pezet D, Bonnet R. High prevalence of mucosa-associated E. coli producing cyclomodulin and genotoxin in colon cancer. PLoS One. 2013;8(2):e56964. doi: 10.1371/journal.pone.0056964. Epub 2013 Feb 14. PMID 23457644
- [Background] Roy S, Trinchieri G. Microbiota: a key orchestrator of cancer therapy. Nat Rev Cancer. 2017 May;17(5):271-285. doi: 10.1038/nrc.2017.13. Epub 2017 Mar 17. PMID 28303904
- [Background] Villeger R, Lopes A, Veziant J, Gagniere J, Barnich N, Billard E, Boucher D, Bonnet M. Microbial markers in colorectal cancer detection and/or prognosis. World J Gastroenterol. 2018 Jun 14;24(22):2327-2347. doi: 10.3748/wjg.v24.i22.2327. PMID 29904241
- [Derived] Taoum C, Carrier G, Jarlier M, Roche G, Gagniere J, Fiess C, De Forges H, Chevarin C, Colombo PE, Barnich N, Rouanet P, Bonnet M. Determination of biomarkers associated with neoadjuvant treatment response focusing on colibactin-producing Escherichia coli in patients with mid or low rectal cancer: a prospective clinical study protocol (MICARE). BMJ Open. 2022 Dec 2;12(12):e061527. doi: 10.1136/bmjopen-2022-061527. PMID 36460331